CLINICAL TRIAL: NCT04377178
Title: Comparison of Autogenous Tooth Graft of Two Different Particle Sizes in Extraction Socket Preservation: A Comparative Clinical and Radiographical Study
Brief Title: Tooth Graft of Two Different Particle Sizes in Extraction Sockets
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: SVS Institute of Dental Sciences (Other)
Responsible Party: Principal Investigator, Dr R Viswa Chandra, Primary Investigator, SVS Institute of Dental Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SVSIDS/PERIO/4/2018
Record Dates: First submitted 2020-04-29; First posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Socket Preservation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dentin chips group from automated mill (Experimental): Dentin particles prepared from dentin grinder will be placed in extraction socket immediately after extraction
  Interventions: Device: Dentin grinder
- Manually milled Dentin chips (Active Comparator): Dentin particles prepared from bone mill will be placed in extraction socket immediately after extraction.
  Interventions: Device: Bone mill

INTERVENTIONS:
Device: Dentin grinder — After atraumatic extraction of the tooth, autogenous dentin particles are made with the help of a device - dentin grinder from the separated root and these particles are incorporated into the extraction socket
  Arms: Dentin chips group from automated mill
Device: Bone mill — After atraumatic extraction of the tooth, autogenous dentin particles are made with the help of a device - Bone mill from the separated root and these particles are incorporated into the extraction socket
  Arms: Manually milled Dentin chips

SUMMARY:
The primary objective of the present study is to clinically and radiographically evaluate the efficacy of autogenous tooth graft obtained from bone mill and dental grinder to preserve alveolar ridge dimensions in extraction sockets.

DETAILED DESCRIPTION:
Accordingly, teeth will be used as a test material to allow for comparative tests after processing it in the automated milling system (AMS). The material will be moistened and then placed in toto into the extraction sockets to generate particles at settings 1 (500 RPM for 30s) or 2 (900 RPM for 30s) to generate MS and SS respectively ((SS group; 0.5-0.8 mm) and medium size (MS group; 1.0-1.2 mm)).

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy individuals within the age group of 20-50 years with presence of teeth with hopeless prognosis requiring extraction

Exclusion Criteria:

* Medically compromised patients.
* Subjects who underwent radiotherapy or chemotherapy in the past 12 months.
* Patients having uncontrolled periodontal disease or having an active sinus infection.
* Smokers

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-05-25 (Actual); Primary Completion 2020-09-25 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Bone fill | Baseline to 6months
  The radiograph obtained at 3 and 6 months will be subtracted from the radiograph taken at the baseline by using commercially available image processing software (Adobe Photoshop® 6.0, Adobe Systems, San Jose, USA). After digital subtraction, the digitized and excluded residual bone height will be transferred to open source software for area calculation (ImageJ®, Research Services Branch, NIH, Bethesda, Maryland, USA) for area calculation. The area of the layer will be calculated (in mm2) by initially enclosing the entire area with the rectangular selection tool and then by using Analyze>Analyze Particles tool.
Bone density | Baseline to 6months
  Radiographs will be taken with digitalized RVG machine (DX 3000, DEXCOWN portable dental X-ray system) at 60Kvp/2Ma with inactive interface. RVG images taken at baseline and 6 months will be utilized to evaluate bone mineral density through Hounsfield units (HU).

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - R V Chandra, Hyderabad, Telangana
  - Svs Institute of Dental Sciences, Hyderabad, Telangana

IPD SHARING:
Plan to Share IPD: No